CLINICAL TRIAL: NCT06130761
Title: Pericapsular Nerve Group Block Combined Versus Trans Muscular Quadratus Lumborum Block in Pediatric Patients Undergoing Correction of Dysplasia of the Hip: a Prospective Randomized Double Blinded Study
Brief Title: Pericapsular Block Versus Trans Muscular Quadratus Lumborum Block in Patients Undergoing Correction of Hip Dysplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aliaa Helmy Mohammed Mohammed, Assistant Lecturer of Anesthesiology, Surgical ICU and Pain management, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MD-302-2022
Record Dates: First submitted 2023-04-09; First posted 2023-11-14 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2023-11

CONDITIONS: Hip Dysplasia
Keywords: quadratus lumborum blocks
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PENG block (P group) (Experimental): PENG BLOCK : 0.5 ml/kg of 0.25% bupivacaine is deposited between the psoas tendon anteriorly and pubic ramus posteriorly lifting it , and to perform the LFCN block 0.1 ml/kg of 0.25% bupivacaine is injected in lateral to femoral artery below anterior superior iliac spine .
  Interventions: Procedure: Pericapsular Nerve Group Block Combined With Lateral Femoral Cutaneous Nerve Block
- TQL block (Q group) (Experimental): QL is usually identified medial to the aponeurosis of transversus abdominis muscle vertically attached above the iliac crest. A 22-gauge 50 mm needle will be inserted in the plane from the posterior edge of the convex probe through the QL in an anteromedial direction. The needle tip will be placed between the PM muscle and the QL muscle and the local anesthetic will be injected into the fascial plane after aspiration test is negative. A volume 0.5 ml/kg of 0.25% bupivacaine is injected with maximum dose 2.5mg per kg of bupivacaine
  Interventions: Procedure: trans muscular quadratus lumborum block

INTERVENTIONS:
Procedure: Pericapsular Nerve Group Block Combined With Lateral Femoral Cutaneous Nerve Block — For PENG block transducer is placed in the transverse plane over the anterior inferior iliac spine (AIIS) and moved inferiorly to visualize the pubic ramus. The femoral artery and iliopubic eminence are visualized, and then, using an in-plane technique, a 22-gauge 50 mm needle is advanced from lateral to medial then 0.5 ml/kg of 0.25% bupivacaine is deposited between the psoas tendon anteriorly and pubic ramus posteriorly lifting it.
  For LFCN the transducer is placed immediately inferior to the anterior superior iliac spine (ASIS), parallel to the inguinal ligament. The tensor fasciae lata muscle (TFLM) and sartorius muscle (SaM) are then identified. The nerve appears as a small hypoechoic oval structure with a hyperechoic rim between the TFLM and SaM in a short-axis view or superficial to the SaM. A 22-gauge 50 mm needle is inserted in-plane in a lateral-to-medial orientation through the subcutaneous tissue. A fascial "pop" may be felt as the needle tip enters the plane.
  Other Names: PENG block
  Arms: PENG block (P group)
Procedure: trans muscular quadratus lumborum block — With the patient in the lateral position, after standard sterilization of skin and probe identify 3 layers of the abdomen. The transversus abdominis is traced more posteriorly until the transversus aponeurosis. usually we can find the peritoneum curves away from the muscles from anterior to posterior . Tilting the probe slightly caudal into the pelvis thus improves the view of the retroperitoneal fat and the tapered end of transversus aponeurosis. QL is usually identified medial to the aponeurosis of transversus abdominis muscle vertically attached above the iliac crest. A 22-gauge 50 mm needle will be inserted in the plane from the posterior edge of the convex probe through the QL in an anteromedial direction. The needle tip will be placed between the PM muscle and the QL muscle and the local anesthetic will be injected into the fascial plane after aspiration test is negative. A volume 0.5 ml/kg of 0.25% bupivacaine is injected with maximum dose 2.5mg per kg of bupivacaine.
  Other Names: TQL block
  Arms: TQL block (Q group)

SUMMARY:
The aim of our study to compare the analgesic effect of pericapsular nerve group block combined with lateral femoral cutaneous nerve block and trans muscular quadratus Lumborum Block block perioperatively in pediatric patients undergoing developmental dysplasia of the hip surgical repair

DETAILED DESCRIPTION:
Patients of both study groups will be monitored using standard monitors Electrocardiogram, pulse oximeter and automated non-invasive blood pressure (NIBP). After preoxygenation, general anesthesia will be induced by a face mask and 8% sevoflurane and 100 % oxygen, then intravenous cannula will be inserted. Fentanyl 1 µg/kg will be given and after neuromuscular block is achieved with atracurium 0.5 mg/kg and the trachea is intubated. Anesthesia will be maintained with isoflurane 1.2% and 60% oxygen and the maintenance dose of atracurium 0.1 mg/kg each 20 minutes. Ringer lactate will be infused at 10 ml/kg per hour in first hour then by the rule 4-2-1 ml per kg per hour.

The blocks will be performed after induction of anesthesia and under ultrasound guidance using SonoSite M Turbo (USA); the scanning probe will be the linear multi-frequency 6-13 MHz transducer (L25 x 6-13 MHz linear array).

Patients will be randomly allocated into two equal groups: PENG block (P group) and TQL block (Q group).

In PENG block group:

With the patient in the supine position, the skin is disinfected, sterile drapes are used, the transducer is wrapped with a sterile dressing, and sterile ultrasound gel is used for scanning, the transducer is placed in the transverse plane over the anterior inferior iliac spine (AIIS) and moved inferiorly to visualize the pubic ramus. The femoral artery and iliopubic eminence are visualized, and then, using an in-plane technique, a 22-gauge 50 mm needle is advanced from lateral to medial through the skin wheal at a 30-degree to 45-degree angle toward the ultrasound beam, Aspiration will be performed before injection, then 0.5 ml/kg of 0.25% bupivacaine is deposited between the psoas tendon anteriorly and pubic ramus posteriorly lifting it .16 To perform the LFCN block: again, the patient in supine position, the skin is disinfected, sterile drapes are used, the transducer is wrapped with a sterile dressing, and sterile ultrasound gel is used for scanning, the transducer is placed immediately inferior to the anterior superior iliac spine (ASIS), parallel to the inguinal ligament. The tensor fasciae lata muscle (TFLM) and sartorius muscle (SaM) are then identified. The nerve should appear as a small hypoechoic oval structure with a hyperechoic rim between the TFLM and SaM in a short-axis view or superficial to the SaM. A 22-gauge 50 mm needle is inserted in-plane in a lateral-to-medial orientation through the subcutaneous tissue. A fascial "pop" or "click" may be felt as the needle tip enters the plane between the TFLM and SaM. To identify the needle tip position, a volume of 0.5-1 mL of isotonic saline may be injected. The correct position is achieved by visualizing the spread of 0.1 ml/kg of 0.25% bupivacaine in the described plane between the TFLM and SaM or around the LFCN superficial to the SaM.9 The dose of bupivacaine in both blocks should not exceed 2.5mg per kg as they will be administrated in the same patient.

In TQL block group:

With the patient in the lateral position, the skin is disinfected, sterile drapes are used, the transducer is wrapped with a sterile dressing, and sterile ultrasound gel is used for scanning, the probe is used to recognize the three layers of abdominal wall muscles. The transversus abdominis is traced more posteriorly until the transversus aponeurosis appears. At this region, usually we can find the peritoneum curves away from the muscles from anterior to posterior and the retroperitoneal fat is visualized. Tilting the probe slightly caudal into the pelvis thus improves the view of the retroperitoneal fat and the tapered end of transversus aponeurosis. QL is usually identified medial to the aponeurosis of transversus abdominis muscle vertically attached above the iliac crest. A 22-gauge 50 mm needle will be inserted in the plane from the posterior edge of the convex probe through the QL in an anteromedial direction. The needle tip will be placed between the PM muscle and the QL muscle and the local anesthetic will be injected into the fascial plane after aspiration test is negative. A volume 0.5 ml/kg of 0.25% bupivacaine is injected with maximum dose 2.5mg per kg of bupivacaine.

In both groups The surgical stimulus will be delayed 15 minutes in both groups. Intraoperative hemodynamics will be recorded at 10minute intervals. If heart rate (HR) increases more than 20% an additional dose of fentanyl 1 µg/kg will be given.

By the end of surgery, inhalational anesthesia will be discontinued and muscle relaxation will be reversed by atropine (0.02 mg/Kg) and neostigmine (0.05 mg/Kg) after the restoration of the patient's spontaneous breathing. The patient will be transferred to the post-anesthesia care unit (PACU) for 2 hours to complete recovery and monitoring. Quality of analgesia will be assessed using (face, legs, activity, and cry consolability scale) (FLACC) pain score18 on admission to PACU and then every 15 minutes for 2 hours. After transfer to the ward, FLACC pain score will be recorded at 3, 6, 12, and 24 hours postoperative.

All patients will receive postoperative diclofenac sodium suppositories 1 mg/kg approximated to available form 12.5 or 25 mg suppository every 8 hours. Morphine IV will be given as rescue analgesia (0.05 mg/kg) in all study groups; if the FLACC pain score (Table 1) is more than 4, the maximum allowed dose will be 0.1mg/kg every 4 hours.

Any complications resulting from peripheral nerve blockade, like local anesthetic systemic toxicity, bleeding, infection or neuropathy, will be recorded and managed accordingly.

ELIGIBILITY:
Inclusion Criteria:

1. Acceptance of the parents
2. Children of both gender
3. ASA I & ASA II
4. Age ranging between 6 months up to 6years old (neglected cases)
5. Scheduled to DDH surgical repair (open reduction or osteotomy) either unilateral or bilateral.
6. Revision cases.

Exclusion Criteria:

1. Parent refusal
2. ASA III, IV
3. Infection at site of block
4. History of allergy to local anesthetics
5. Bleeding disorders with INR > 1.5 and/or platelets < 100,000/mm3

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Time to first rescue analgesia . | 15 minutes after extubation for 24 hours postoperative
  Time to first rescue analgesia 15 minutes after extubating the patient .

SECONDARY OUTCOMES:
Postoperative (FLACC)Face, Legs, Activity, Cry, Consolability scale. | 15 minutes after extubation for 24 hours postoperative
  Postoperative FLACC pain scores with 0 minimum pain and 10 maximum pain
Total intraoperative analgesic (fentanyl) requirements | Intraoperative
  Total amount of analgesics given intraoperative
Total postoperative analgesic requirements | 15 minutes after extubation for 24 hours postoperative
  Total amount of analgesics given postoperative
Intraoperative hemodynamics every 10minutes heart rate, systolic, diastolic, mean arterial blood pressure | Intraoperative
  measuring and recording vitals every 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesia Department, Kasralainy Faculty of Medicine, Cairo University., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No